CLINICAL TRIAL: NCT04713085
Title: Sacral Neuromodulation for Constipation and Fecal Incontinence in Children and Adolescents - Randomized Controlled Trial on the Application of Invasive vs. Non-invasive Technique
Brief Title: Sacral Neuromodulation in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Dr. med. Sonja Diez, Principal Investigator, M.D., Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18_20B2
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Constipation With Overflow; Encopresis With Constipation and Overflow Incontinence; Hirschsprung's Disease; Anorectal Malformations; Sacral Dysgenesis
Keywords: Sacral Nerv Stimulation; Neuromodulation
MeSH Terms: conditions — Hirschsprung Disease; Anorectal Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacral Neuromodulation (Active Comparator): Sacral neuromodulation is surgically implanted within two surgeries:
  1. Implantation of the final electrode (tined-lead electrode): This electrode is implanted to neuronal fibers of S3/4. Both sides are tested intraoperatively, the side with a sufficient response at lower intensity levels is finally implanted. Stimulation is conducted via an external pulse generator.
  2. Implantation of the internal pacemaker system 4 weeks after the electrode's implantation.
  Stimulation parameters: Single current, frequency 15Hz, duration 210μs. Stimulation intensity is individually determined beyond the pain threshold (adjustable amplitude between 0-10mA, depending on the intraoperative response).
  Start point of clinical evaluation is time of implantation of tined lead electrode.
  Medical and behavioral therapy is to be continued as started before intervention.
  Interventions: Device: Invasive Sacral Neuromodulation
- Non-invasive Sacral Neuromodulation (Active Comparator): Two adhesive electrodes are placed paravertebrally between L1 and L4 and periumbilically, generating an electrical field by single current with a 15 Hz frequency for a duration of 210μs. Stimulation intensity is individually determined to achieve an effective and comfortable stimulation beyond the pain threshold (adjustable amplitude between 0-10mA).
  Start point of clinical evaluation is start of external stimulation.
  Medical and behavioral therapy is to be continued as started before intervention.
  Interventions: Device: Non-invasive Sacral Neuromodulation

INTERVENTIONS:
Device: Invasive Sacral Neuromodulation — Internal, implanted sacral nerve stimulation (electrodes in contact with neuronal fibers S3/4)
  Arms: Sacral Neuromodulation
Device: Non-invasive Sacral Neuromodulation — External, non-invasive sacral nerve stimulation via two cutaneously adhesive electrodes (single current).
  Arms: Non-invasive Sacral Neuromodulation

SUMMARY:
The purpose of this study is to assess the efficacy of neuromodulation for treatment of chronic constipation and fecal incontinence in pediatric patients and to evaluate the differences between the invasive vs. non-invasive approach.

DETAILED DESCRIPTION:
Patients are selected according to the eligibility requirements. After obtaining informed consent off-label use and potential risks of sacral neuromodulation, all included patients and next of kin give written informed consent to the study.

At baseline, patients are randomized to one of the two predefined subgroups: either invasive sacral neuromodulation or non-invasive sacral neuromodulation. Clinical symptoms and outcome variables are compared regarding the beginning of non-invasive sacral neuromodulation or the implantation of the tined lead electrode. Patients are closely monitored within 6 months. Treatment success is evaluated in routine clinical check-ups (week 4/8/12 and 24) and via specialized questionnaires and bowel movement diaries. Quality of life is evaluated at baseline and after 12 and 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age between 2-17 years
* informed consent
* chronic constipation according to the ROME IV criteria for more than 3 months with or without encopresis/soiling despite underlying diseases such as slow-transit constipation, rectal evacuation disorders or Hirschsprung's disease.
* refractory to conventional treatment in an appropriate weight-adapted application (training for bowel movements, lifestyle changes, pelvic floor training, pharmacological options)
* in cases of Hirschsprung's disease: diagnosis confirmed histologically by rectal biopsies and in case of resection of an aganglionic segement: period between surgery and SNM at least 1 year
* in cases of anorectal malformation or mechanical obstruction: post-surgical status: period between surgery and SNM at least 1 year

Exclusion Criteria:

* metabolic, inflammatory, and hormonal causes for chronic constipation
* toxic megacolon or further emergencies, which must be treated surgically
* sacral fractures or substantial differences in the sacral anatomy
* inflammatory bowel disorders
* rectal prolapse
* neuronal malignancies under medical and radiation therapy
* seizures

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change of episodes of abdominal pain | Baseline and 12 and 24 weeks after start of therapy
  Abdominal pain is recorded in number of episodes per week. Its intensity is evaluated via the numeric rating scale (0=no pain, 10=worst imaginable pain). Definition of success: reduction by at least 50% of episodes per week
Change of episodes of fecal incontinence | Baseline and 12 and 24 weeks after start of therapy
  Number of episodes of fecal incontinence per week. Definition of success: reduction by at least 50% of episodes per week
Change of defecation frequency | Baseline and 12 and 24 weeks after start of therapy
  Defecation frequency is measured by number of bowel movements per week. Definition of success: doubling of episodes per week to at least 3 or more bowel movements per week
Change of defecation consistency | Baseline and 12 and 24 weeks after start of therapy
  Defecation consistency is measured daily by the Bristol Stool Scale, which classifies stool consistency from 1 (hard consistency) to 7 (fluid consistency). Definition of success: change of at least 2 points within the scale of 1-7

SECONDARY OUTCOMES:
Change of proprioception | Baseline and 12 and 24 weeks after start of therapy
  Improvement of proprioception is measured as mentioned in the specialized questionnaires.
Episodes of urinary incontinence | Baseline and 12 and 24 weeks after start of therapy
  The number of episodes per week is evaluated with the criterion for a clinically relevant improvement in cases of reduction by at least 50% of episodes per week.
Change of Quality of Life | Baseline and 12 and 24 weeks after start of therapy
  The quality of life is classified via the 'Revised Children's Quality of Life Questionnaire' (KINDLR). It consists of 24 5-point Likert-scale items, covering 6 quality of life dimensions: physical well-being, emotional well-being, self-esteem, family, friends and daily functioning (school or nursery school/kindergarten). Items are partially reverse scored and linearly transformed to a 0 to 100 scale according to the manual. Higher scores indicate a better quality of life.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Baseline and 12 and 24 weeks after start of therapy
  Adverse events are measured as mentioned in the specialized questionnaires: these include cutaneous reactions, urinary incontinence, dysfunction of stimulation or further unknown factors.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Diez, M.D., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg; Manuel Besendörfer, M.D., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Friedrich-Alexander-Universität Erlangen-Nürnberg, Pediatric Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Besendorfer M, Kirchgatter A, Carbon R, Weiss C, Muller H, Matzel KE, Diez S. Sacral neuromodulation for constipation and fecal incontinence in children and adolescents - study protocol of a prospective, randomized trial on the application of invasive vs. non-invasive technique. Trials. 2024 Mar 22;25(1):210. doi: 10.1186/s13063-024-08052-6. PMID 38515199